CLINICAL TRIAL: NCT06460441
Title: Comparison of the SUNRISE© Device With Ventilatory Polygraphy for the Diagnosis of Obstructive Sleep Apnea Hypopnea Syndrome: Collection of Preliminary Data
Acronym: SUNPV
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Collaborators: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: GHRMSA 1350
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea Hypopnea Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Suspected OSAHS
  Interventions: Diagnostic Test: SUNRISE© device

INTERVENTIONS:
Diagnostic Test: SUNRISE© device — The device under study is the Sunrise© sensor, a single-use Class IIa medical device with CE marking and ISO 13485 certification.
  The system combines a mandibular movement sensor with an artificial intelligence program to collect and interpret data. It consists of a three-gram device that is placed on the chin using an adhesive. The sensor is linked to a (free) mobile app, enabling data to be sent to the Sunrise© company's secured platform at the end of the night, and results to be transmitted to the prescribing physician.

SUMMARY:
Additional data on screening for obstructive sleep apnea/hypopnea syndrome (OSAHS) in patients with co-morbidities, such as diabetics and those with chronic respiratory diseases would enable current recommendations to evolve, with a view to promoting the widespread use of simplified techniques for OSAHS screening, particularly in patients with cardiorespiratory co-morbidities.

The primary objective of this observational multicentric pilot study is to compare the performance of the Sunrise® medical device with that of ventilatory polygraphy as part of routine screening for OSAHS in diabetic patients followed up in the diabetology department of the Strasbourg University Hospital, and in patients followed up in the pneumology consultation department of Mulhouse Hospital (GHRMSA).

DETAILED DESCRIPTION:
Secondary objectives

1. To assess the correlation of the following parameters:

   * dorsal Apnea-Hypopnea Index (AHI) measured by ventilatory polygraphy and dorsal Obstructive Respiratory Disturbance Index (ORDI) measured by Sunrise® device
   * non-dorsal AHI measured by ventilatory polygraphy and non-dorsal ORDI measured by Sunrise® device
2. To study the correlation between AHI measured by the Sunrise® medical device and desaturation index measured by ventilatory polygraphy.

Conduct of research

* At Strasbourg University Hospital, the study will be proposed to patients admitted for diabetic assessment who require ventilatory polygraphy.
* At Mulhouse hospital (GHRMSA), patients are referred to a pneumologist in case of suspected OSAHS and a ventilatory polygraphy is scheduled at home. Patients scheduled to undergo this examination will be invited to take part in the study.

Ventilatory polygraphy (routine care):

Patients included in the study will receive an additional recording using the Sunrise© medical device, performed simultaneously with the ventilatory polygraphy.

Ventilatory polygraphy will be performed in accordance with each center's usual practices. For patients undergoing home polygraphy (GHRMSA), the care team will install the sensors and program the device for recording during sleep. The patient will return home and spend the night there, before coming back to the hospital the following day to give back the equipment. For patients hospitalized in the diabetology department of Strasbourg University Hospital, ventilatory polygraphy will be carried out during hospitalization.

Sunrise© medical device (examination added by research):

The mobile application will be installed on patient's smartphone by the study investigating team, and the use of the Sunrise© device will be explained to the patient. Recording will take place on the same night as the ventilatory polygraphy.

The day after recording, the Sunrise© sensor and ventilatory polygraph equipment will be collected by the investigating team.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over;
* Patient with a smartphone (Android or iOS) with Bluetooth and Internet connection and able to use the mobile application associated with the Sunrise© medical device;
* Patient having a scheduled exploration by ventilatory polygraphy;
* Non-opposition to participation in the research.

Exclusion Criteria:

* Patient suffering from a psychiatric pathology or with a history of behavioral disorders;
* Patient already treated for OSAHS;
* Patient refusing to cut his beard (if too abundant to wear the Sunrise© device);
* Patient suffering from a pathology affecting the rotation of the condyle in the temporomandibular joint;
* Patient deprived of liberty by judicial or administrative decision;
* Patients under court protection or legal guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be proposed to diabetic patients treated in the diabetology department of the Strasbourg University Hospital, as well as to patients referred to the pneumology consultation at the GHRMSA (Mulhouse) who need to have their sleep disorders investigated using ventilatory polygraphy.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | Day 1
  The apnea-hypopnea index (AHI) will be measured using the Sunrise® medical device and ventilatory polygraphy. It corresponds to the number of apnea-hypopnea episodes per hour of sleep.

SECONDARY OUTCOMES:
Dorsal AHI | Day 1
Non- dorsal AHI | Day 1
Dorsal Obstructive respiratory disturbance index (ORDI) | Day 1
Non dorsal ORDI | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, Bas-Rhin, France

IPD SHARING:
Plan to Share IPD: No